CLINICAL TRIAL: NCT06813807
Title: A Comparative Study of the Pharmacokinetic Profiles of Timolol Maleate Ophthalmic Gel Forming Solution After Multiple Dosing in Healthy Subjects With That of Timolol Maleate Gel in Subjects With Proliferating Superficial Infantile Hemangioma Who Have Completed the Study
Brief Title: A Comparative Study of the Pharmacokinetic Profiles of Timolol Maleate Ophthalmic Gel With Timolol Maleate Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auson Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASN001C003-CN
Record Dates: First submitted 2025-01-23; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 0.5%TM (Experimental): 18 subjects will receive one drop of 0.5% timolol maleate ophthalmic gel forming solution each in the left and right eyes once daily.
  Interventions: Drug: 0.5% TM

INTERVENTIONS:
Drug: 0.5% TM — From D1 to D10, each subject will receive one drop of 0.5% timolol maleate ophthalmic gel forming solution each in the left and right eyes once daily at the same time every day under fasted condition.

SUMMARY:
The goal of this clinical trial is:

1)To evaluate the pharmacokinetic profiles and safety of 0.5% Timolol Maleate Ophthalmic Gel Forming Solution in healthy adult subjects after multiple dosing; 2)To compare the systemic exposure (Cmax,ss and AUCss) of 0.5% Timolol Maleate Gel in subjects with proliferating superficial infantile hemangioma (completed) with that of 0.5% Timolol Maleate Ophthalmic Gel Forming Solution in healthy adult subjects.

The main questions aim to answer are:

* Pharmacokinetic (PK) profiles of healthy adult subjects
* Safety Evaluation
* To compare the systemic exposure (Cmax,ss and AUCss) of 0.5% timolol maleate gel in subjects with proliferating superficial infantile hemangioma (completed) with that of 0.5% timolol maleate ophthalmic gel forming solution in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: Healthy male or female subjects aged 18 to 50 years old (inclusive);
2. Weight: ≥ 50 kg for male, ≥ 45 kg for female; body mass index (BMI) between 19 and 26 kg/m2 (inclusive), where BMI = weight (kg) / height2 (m2);
3. Ophthalmic examinations during screening include visual acuity, color vision, intraocular pressure, slit-lamp examination (of eyelids, lacrimal apparatus, anterior chamber, conjunctiva, etc.) and fundus examination must be normal or abnormal without clinical significance;
4. Refractive myopia < 600 degrees, corrected visual acuity ≥ 0.8 in both eyes;
5. Subjects with no abnormal or with abnormal but not clinically significant results in vital signs measurement, physical examination, clinical laboratory tests (hematology, urinalysis, blood biochemistry, infectious disease test and coagulation function), pregnancy test (women of childbearing age), and 12-lead ECG;
6. Male subjects and their partners or female subjects must agree to take one or more non-drug contraceptive measures (such as complete abstinence, intrauterine ring and partner ligation) during the study and for 3 months after the end of the study, and have no plan of sperm or egg donation; Subjects have a full understanding of the study content, investigational drugs, study process, etc., and are able to communicate well with the investigator, willing to comply with the study regulations, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. (Screening period inquiry + check-in inquiry) Subjects with a history of respiratory system (especially bronchial asthma, bronchospasm, chronic obstructive pulmonary disease), cardiovascular system, digestive system, endocrine system, urinary system, nervous system, hematological, immunological, psychiatric disorders or a family history of genetic psychosis, cancer, etc., and are considered by the investigator to still have clinical significance;
2. (Screening period inquiry) Subjects with a history of diabetes, thyrotoxicosis, cardiogenic shock, second- to third-degree atrioventricular block, heart failure, significant sinus bradycardia, hypotension, sick sinus syndrome, severe peripheral vascular disease with resting ischemia and whose condition is assessed by the study physician to be abnormal but clinically significant;
3. (Screening period inquiry + check-in inquiry) Subjects who have undergone surgery within 6 months before the first dose that will affect drug absorption, distribution, metabolism and excretion as judged by the investigator; or who have undergone surgery within 4 weeks before the first dose; or who plan to undergo surgery during the study period;
4. (Screening period inquiry) Subjects with a history of or currently suffering from any acute and chronic eye diseases, or with ocular mixed infections, inflammation, trauma or other ophthalmic conditions with clinical significance(e.g., keratoconus, severe dry eye) within 1 month before the first dose, active eye diseases, or acute or chronic allergic eye diseases or any abnormalities in the eyelids, ocular surface, and lacrimal passage system that may affect the absorption of eye drops in the opinion of the investigator;
5. (Screening period inquiry) Subjects with a history of ocular trauma or eye surgery;
6. Subjects whose elevated intraocular pressure exceeds the normal range (10 ~ 21 mmHg), with the pressure difference of greater than 5 mmHg between both eyes and considered clinically significant by the study doctor;
7. Subjects with keratopathy, corneal thickness greater than 600 um (normal central corneal thickness is 500 ~ 600 um) or corneal scarring, wearing contact lenses (including night wear orthokeratology lenses) or having to wear contact lenses during the study, which affect the intraocular pressure measurement and are considered clinically significant by the study physician;
8. (Screening period inquiry) Those with evidence or a history of acute and chronic angle-closure glaucoma;
9. (Screening period inquiry + check-in inquiry) Those who have used any drugs that inhibit or induce hepatic drug metabolizing enzymes or interact with the study drugs (adrenoceptor inhibitors, digitalis and calcium antagonists, catecholamine-depleting drugs, clonidine, quinidine, etc.) within 30 days prior to the first dose;
10. (Screening period inquiry + check-in inquiry) Subjects who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, vaccines or health products for various reasons within 14 days prior to the first dose in the study;
11. (Screening period inquiry) Subjects who are allergic to timolol maleate ophthalmic gel forming solution or its excipients; or those who are allergic to two or more items of other drugs, foods and environment; or those with allergic constitution who are prone to allergic symptoms such as rash (generalized rash, urticaria) and itching;
12. (Screening period inquiry + check-in inquiry) Individuals with a history of drug abuse, drug dependence or positive results of drug abuse screening (morphine, methylamphetamine, ketamine, methylenedioxymethamphetamine, tetrahydrocannabinolic acid, cocaine);
13. (Screening period inquiry + check-in inquiry) Those who are former smokers or have smoked more than 5 cigarettes per day on average within 3 months before screening, or are unable to stop using any tobacco products during the study;
14. (Screening period inquiry + check-in inquiry) Subjects with a history of alcoholism/alcohol abuse or who are regular drinkers within 6 months prior to screening (ie, consuming more than 14 standard units of alcohol per week, where 1 standard unit equals to 17.5 mL or 14 g of pure alcohol. Alcohol content of different types of alcoholic beverages is indicated by volume ratio, 1 standard unit approximately equals to 35 mL of 50° liquor or 350 mL of 5° beer), or those who are unwilling to stop drinking or consuming any alcohol-containing products during the study, or with alcohol breath test results > 0.0 mg/100 mL;
15. (Screening period inquiry + check-in inquiry) Subjects who have previously consumed excessive amounts of tea, coffee and/or caffeine-rich, grapefruit, xanthine-rich beverages (including tea, caffeine, cocoa) for a long period of time (more than 8 cups per day on average, 1 cup = 200 mL), or who have consumed any caffeine-rich, grapefruit-rich beverages or foods within 7 days before the first dose, or who do not agree to stop eating the above diet during the study;
16. (Screening period inquiry) Subjects who have special requirements for diet and cannot follow the standardized diet of the site;
17. (Screening period inquiry + check-in inquiry) Those who have donated or lost a large amount (≥ 400 mL) of blood within 3 months prior to enrollment or plan to donate blood or blood components within 3 months after the end of the study;
18. (Screening period inquiry + online screening) Subjects who have participated in any clinical study and used the investigational drug within 90 days before screening;
19. (Screening period inquiry) Subjects with a history of fainting due to needles or blood, difficulty in venous blood sampling and/or intolerance to venipuncture/indwelling needle;
20. Subjects who have skin damage or scars or skin diseases at the application site (around the eyes) and cannot be enrolled at the investigator's discretion; Other factors that, in the opinion of the investigator, make the subject unsuitable for participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | 24 hours after administration
  maximum plasma concentration at steady state
AUC0-t,ss | 24 hours after administration
  area under the plasma concentration-time curve from the last dose to the collection time t of the last measurable concentration
AUC0-24,ss | 24 hours after administration
  area under the plasma concentration-time curve over a 24-h dosing interval at steady state
AUC0-∞,ss | 24 hours after administration
  area under the plasma concentration-time curve extrapolated from the last dose to infinity at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Huzhou Central Hospital, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No